CLINICAL TRIAL: NCT05996146
Title: Incidence of Hoarseness After General Spine Surgery: Prospective Observational Study
Acronym: Hoarseness
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Clinical Professor, Seoul National University Hospital
Other Study IDs: HA-427
Record Dates: First submitted 2023-07-24; First posted 2023-08-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hoarseness
Keywords: hoarseness; spine surgery
MeSH Terms: conditions — Hoarseness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hoarseness group: This study recruited all patients admitted at Seoul National University Hospital.
  Age range is 20 to 80 years old. Patients who require surgical treatment for degenerative spine conditions. Patients who voluntarily consent to participate in the study.

SUMMARY:
Early diagnosis and appropriate treatment of hoarseness is known to improve quality of life and treatment outcomes. Therefore, appropriate research on the incidence of hoarseness after surgery is necessary. In this study, investigator aim to investigate incidence of hoarseness after spine surgery and the correlation between the Voice Handicap Index (VHI)-10, used as a criterion, and acoustic parameters, while also validating the efficacy of our research methods.

DETAILED DESCRIPTION:
The primary outcome of this study is the incidence of hoarseness on the day of surgery.

The secondary outcomes include the incidence of hoarseness at one month after surgery, as well as examining the correlation between acoustic parameters, risk factors, and the occurrence of hoarseness.

Investigator conducted a comparative analysis of risk factor for hoarseness in patients with different VHI-10 scores on the day of surgery and 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age range is 20 to 80 years old
* degenerative spine conditions
* visit at Seoul National University Hospital only
* Patients who voluntarily consent to participate in the study

Exclusion Criteria:

* History of surgery around the airway or mediastinum
* patients with vocal cord-related disorders
* Patients with fractures, bleeding, or other trauma
* Patients with neuromuscular diseases, Parkinson's disease, or psychiatric disorders
* Patients who cannot be extubated or who are transferred to the ICU after surgery
* Pregnant women
* Patients who do not wish to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age range is 20 to 80 years old. Patients who require surgical treatment for degenerative spine conditions and visit at Seoul National University Hospital. Patients who voluntarily consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
the primary outcome was to measure the incidence of hoarseness | voice recordings six hours after the end of anesthesia
  the primary outcome was to measure the incidence of voice disorders by conducting Voice Handicap Index-10 (minimum score 0 to maximum score 46, lower score is better) scoring and voice recordings six hours after the end of anesthesia

SECONDARY OUTCOMES:
The secondary outcome involved measuring the incidence of hoarseness one month after the surgery | one month after the surgery
  analyzed the correlation between Voice Handicap Index-10 (minimum score 0 to maximum score 46, lower score is better) scores and voice acoustic parameter analysis

CONTACTS AND LOCATIONS:
Overall Officials: SUM KIM, Dr, Principal Investigator — Department of Neurosurgery, Seoul National University Hospital, Republic of Korea.
Locations (1):
- Seoul National University Hospital, Seoul, South Korea